CLINICAL TRIAL: NCT04173377
Title: Elbow Outcomes Clinical Study (WELBOW)
Acronym: WELBOW
Status: Completed | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: 1801-T-WELBOW-RM; 2019-A00492-55 (Other: French National Health Agency)
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Orthopedic Disorder
Keywords: Orthopedic Surgery; Elbow; Trauma; Arthroplasty; Osteosynthesis
MeSH Terms: conditions — Musculoskeletal Diseases; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
WELBOW study is an international, ambispective and prospective, single arm, multicenter, observational, non-comparative, Post-Market Clinical Follow-up (PMCF).

DETAILED DESCRIPTION:
WELBOW study is an international, ambispective and prospective, single arm, multicenter, observational, non-comparative, Post-Market Clinical Follow-up (PMCF). Outcome data collected from this study will provide the basis for Post-Market Surveillance (PMS) reporting, Clinical Study Report (CSR) and Clinical Evaluation Report (CER) on Elbow system devices and support peer-reviewed publications on long-term product performance and safety.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of the informed consent or the non-opposition (when applicable).
* Informed and willing to sign an informed consent form approved by IRB or EC (when applicable).
* Willing and able to comply with the requirements of the study protocol.
* For prospective inclusion: Considered for treatment with one Wright Medical Elbow arthroplasty or fracture devices included in this study (primary or revision).
* For ambispective inclusion

  1. Must have undergone an Elbow arthroplasty or fracture with one Wright Medical Elbow studied device between the date of the first Site Initiation Visit (SIV) and until 4.5 years prior this one in order to have at least the 5 years follow-up visit prospectively. Ambispective patients who were explanted prior the date of the first SIV will be included.
  2. Must have complete Information available for each completed visit (demographics, preoperative information, surgery information, device details)*.

Exclusion Criteria:

* Not able to comply with the study procedures based on the judgment of the assessor (e.g. cannot comprehend study questions, inability to keep scheduled assessment times).
* Patient belongs to a vulnerable group of patients, including minor patients, those unable to decide for themselves to participate or needing a Legally Authorized Representative (LAR), or others who could be subject to coercion (patients who may not be acting on their own initiative) (referred as "vulnerable subject" in the section 3.44 of the ISO 14155:2011 norm).
* Patient with previous elbow device(s) which remain(s) implanted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Europe (United Kingdom, France, Germany, Sweden, Belgium) and Canada
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Clinical Assessment: QuickDASH questionnaire | At 24 months
  Demonstrate a superior (lower) Total QuickDASH score average at 24 months postoperative compared to the upper threshold of 49 points The QuickDASH is an abbreviated 11-question subset from the original Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire. The questionnaire's answers are scored on a 1-5 points scale that is then transformed to result in a score that ranges from 0 (indicating least disability) to 100 (indicating most disability).

SECONDARY OUTCOMES:
Safety and Tolerability : Number of device associated and procedure associated adverse events. | Up to 10 years.
  Number of device associated and procedure associated adverse events.
Implant Survivorship | At 2, 5, 7 and 10 years.
  Rates of revision surgeries; assessed using the Kaplan-Meyer analysis. Censorship will be at the point of the last patient event (visit, death, revision).
Clinical Assessment: MEPS questionnaire | From Baseline to 10 years except 7 years.
  Clinician based index with 4 subscales and 8 items (pain, range of motion, stability, daily function), measured with a goniometer. MEPS ranges from 5 to 100 points which higher scores indicates better function. A total score between 90 and 100 points considered excellent; between 75 and 89 points, good; between 60 and 74 points; fair, less than 60 points, poor
Clinical Assessment: QuickDASH questionnaire | From Baseline to 10 years except 7 years.
  The QuickDASH is an abbreviated 11-question subset from the original Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire. The questionnaire's answers are scored on a 1-5 points scale that is then transformed to result in a score that ranges from 0 (indicating least disability) to 100 (indicating most disability).
Clinical Assessment: Range of Motion | From Baseline to 10 years except 7 years.
  Range of Motion (ROM) is a movement test conducted on a joint to diagnose level of pain and function. Flexion / Extension, Supination and Pronation will be evaluated.
Clinical Assessment: Strength | From Baseline to 10 years except 7 years.
  Elbow strength will be measured with the MRC Strenght Scale The MRC Strength Scale is a 5-items scale. The muscle scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle. Grade 5 shows normal contraction of the muscle, Grade 0 shows no movement.
Clinical Assessment: Patient's Satisfaction | From Baseline to 10 years except 7 years.
  * Single subjective question: "How satisfied are you with your elbow?" Response options include: "Very Satisfied, Satisfied, Dissatisfied, and Very Dissatisfied".
  * Subjective value: "How would you rate your elbow today as a percentage of normal? (0 to 100% scale with 100% being normal)".
Radiologic Assessment for bone characteristics | Before surgery, at 3 months for Osteosynthesis and 1, 2, 5 and 10 years for Arthroplasties.
  Imaging (X-ray, CT scan or MRI) will be analyzed, when sufficient information is available, for bone characteristics
Radiologic Assessment for device migration | Before surgery, at 3 months for Osteosynthesis and 1, 2, 5 and 10 years for Arthroplasties.
  Imaging (X-ray, CT scan or MRI) will be analyzed, when sufficient information is available, for device migration

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma
Locations (7):
- AZ Herentals, Herentals, Belgium
- Lawson Health Research Institute, London, Canada
- France (4):
  - CHU Bordeaux, Bordeaux
  - Clinique du parc, Lyon
  - CHU de Rouen, Rouen
  - CHU Tours, Tours
- Wrightington Hospital, Wigan, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No